CLINICAL TRIAL: NCT01249404
Title: A Phase III, Multicentre, Double-blind, Prospective, Randomized, Placebo-controlled Study, Assessing the Efficacy and Safety of Dysport® Used for the Treatment of Lower-limb Spasticity in Adult Subjects With Hemiparesis Due to Stroke or Traumatic Brain Injury
Brief Title: Dysport® Adult Lower Limb Spasticity Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Y-55-52120-140; 2009-015868-34 (EudraCT Number)
Record Dates: First submitted 2010-11-25; First posted 2010-11-29 (Estimated); Results first posted 2017-10-17 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Leg Spasticity
MeSH Terms: interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dysport® 1000 U, IM (Experimental): 1000 U, I.M. (in the muscle), on day 1 (single treatment cycle)
  Interventions: Biological: Botulinum toxin type A
- Dysport® 1500 U, IM (Experimental): 1500 U, I.M., on day 1 (single treatment cycle)
  Interventions: Biological: Botulinum toxin type A
- Placebo (Placebo Comparator): I.M., on day 1 (single treatment cycle)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Botulinum toxin type A — I.M. injection on day 1 (single treatment cycle)
  Other Names: AbobotulinumtoxinA (Dysport®)
  Arms: Dysport® 1000 U, IM; Dysport® 1500 U, IM
Drug: Placebo — I.M. injection on day 1 (single treatment cycle)
  Arms: Placebo

SUMMARY:
The purpose of this research study is to assess the efficacy of Dysport® compared to placebo in improving muscle tone in hemiparetic subjects with lower limb spasticity due to stroke or traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 to 80 years of age
* Post stroke or brain injury
* Intensity of muscle tone greater than or equal to 2, as measured on the Modified Ashworth Scale
* Ambulatory patients

Exclusion Criteria:

* Fixed contractures
* Physiotherapy initiated less than 4 weeks before entry
* Previous surgery or previous treatment with phenol and/or alcohol in lower limb
* Neurological/neuromuscular disorders which may interfere with protocol evaluations

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Study Director, Study Director — Ipsen
Locations (62):
- United States (17):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Rancho Los Amigos, Downey, California
  - Pacific Neuroscience Medical Group, Oxnard, California
  - Associated Neurologists of Southern CT, PC, Fairfield, Connecticut
  - Parkinson's Disease & Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Design Neuroscience, Miami Gardens, Florida
  - Mount Sinai School of Medicine, New York, New York
  - Weill Cornell Medical College, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - MossRehab & Albert Einstein, Elkins Park, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - The University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of North Texas HSC at Ben Hogan Center, Fort Worth, Texas
  - Neurorehabilitation Specialist, Houston, Texas
  - University of Texas - Houston, Houston, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
- Australia (8):
  - Epworth HealthCare, Richmond, Victoria
  - Caulfield Hospital, Caulfield
  - Saint Vincent's Hospital, Darlinghurst
  - Saint Vincent's Hospital, Fitzroy
  - St George Hospital, Kogarah
  - Royal Melbourne Hospital, Parkville
  - Epworth Healthcare, Richmond
  - Westmead Hospital, Westmead
- Belgium (2):
  - Université catholique de Louvain av Hippocrate 10, Brussels
  - Clinique Universitaire, Yvoir
- Czechia (2):
  - Neurologicka Klinika, Olomouc
  - Neurologicka Klinika, VFN, Prague
- France (10):
  - CHU Jean MINJOZ, Besançon
  - Service de Réeducation Fonctionnelle, CHU de Brest, Hôpital Morvan, Brest
  - Centre de Réadaptation de Coubert, Coubert
  - Centre Hospitalier Albert Chenevier, Créteil
  - Hopital Raymond Poincarré, Garches
  - Hôpital de L'Archet, Nice
  - Hôpital Sébastopol, Médecine Physique et Réadaptation, CHU Reims, Reims
  - Hôpital Sébastopol, Reims
  - Nouvel Civil Hospital, Strasbourg
  - Hopital Rangueil, Toulouse
- Hungary (5):
  - National Institute for Medical Rehabilitation, Budapest
  - Szent János Hospital, Budapest
  - Uno Medical Trials, Budapest
  - Petz Aladar Country Hospital, Győr
  - Batthyány Kázmér Hospital, Kisbér
- Italy (4):
  - Azienda Ospedaliero, Catania
  - SSD Neurofisiologia Riabilitativa, Fossano
  - Servizio di Neurofisiologia Clinica-Ospedale San Raffaele, Milan
  - Polo IRCCS Eugenio Medea La Nostra Famiglia, Treviso
- Poland (6):
  - Specjalistyczna Praktyka Lekarska, Katowice
  - Centrum Medyczne Plejady, Krakow
  - Krakowska Akademia Neurologii, Krakow
  - Malopolskie Centrum Medyczne, Krakow
  - Nzoz Neuro - Card, Poznan
  - Samodzielny Publiczny Centralny Szpital, Warsaw
- Portugal (3):
  - Servicio de Rehabilitation de Adultos, Alcabideche
  - Centro Hospitalar Lisboa Norte, Lisbon
  - Centro Hospitalar São João, Porto
- Russia (3):
  - Treatments and Rehabilitation Center, Moscow
  - State Institution "Scientific Centre of Neurology of Russian Academy of Medical Sciences", Saint Petersburg
  - St-Petersberg State Medical University, Saint Petersburg
- Slovakia (2):
  - Neurologicka klinika, Univerzitna nemocnica Bratislava, Bratislava
  - Univerzitna Nemocnica Bratislava, Bratislava

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Derived] Esquenazi A, Brashear A, Deltombe T, Rudzinska-Bar M, Krawczyk M, Skoromets A, O'Dell MW, Grandoulier AS, Vilain C, Picaut P, Gracies JM. The Effect of Repeated abobotulinumtoxinA (Dysport(R)) Injections on Walking Velocity in Persons with Spastic Hemiparesis Caused by Stroke or Traumatic Brain Injury. PM R. 2021 May;13(5):488-495. doi: 10.1002/pmrj.12459. Epub 2020 Sep 11. PMID 32741133
- [Derived] Esquenazi A, Stoquart G, Hedera P, Jacinto LJ, Dimanico U, Constant-Boyer F, Brashear A, Grandoulier AS, Vilain C, Picaut P, Gracies JM. Efficacy and Safety of AbobotulinumtoxinA for the Treatment of Hemiparesis in Adults with Lower Limb Spasticity Previously Treated With Other Botulinum Toxins: A Secondary Analysis of a Randomized Controlled Trial. PM R. 2020 Sep;12(9):853-860. doi: 10.1002/pmrj.12348. Epub 2020 Mar 27. PMID 32108436
- [Derived] Gracies JM, Esquenazi A, Brashear A, Banach M, Kocer S, Jech R, Khatkova S, Benetin J, Vecchio M, McAllister P, Ilkowski J, Ochudlo S, Catus F, Grandoulier AS, Vilain C, Picaut P; International AbobotulinumtoxinA Adult Lower Limb Spasticity Study Group. Efficacy and safety of abobotulinumtoxinA in spastic lower limb: Randomized trial and extension. Neurology. 2017 Nov 28;89(22):2245-2253. doi: 10.1212/WNL.0000000000004687. Epub 2017 Nov 1. PMID 29093068

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was designed as a mutlicentre study and included 62 investigational centres in Australia, Belgium, the Czech Republic, France, Hungary, Italy, Poland, Portugal, Russia, Slovakia and the United States. Subjects were screened at 53 centres and in 52 centres subjects were randomised to receive study treatment.
Pre-assignment Details: A total of 456 subjects were screened, 388 were enrolled into the study and randomised to 1 of 3 treatment groups.
Groups:
- Dysport® 1000 U: Subjects received intramuscular (i.m.) injections of Dysport® 1000 Units (U) (maximum total dose) into the soleus muscle and gastrocnemius (medial and/or lateral) muscle and at least one of the distal or proximal muscles of the leg on Day 1 of the single treatment cycle. Dysport® contains the neurotoxin Clostridium botulinum type A toxin-haemagglutinin complex (abobotulinumtoxinA).
- Dysport® 1500 U: Subjects received i.m. injections of Dysport® 1500 U (maximum total dose) into the soleus muscle and gastrocnemius (medial and/or lateral) muscle and at least one of the distal or proximal muscles of the leg on Day 1 of the single treatment cycle. Dysport® contains the neurotoxin Clostridium botulinum type A toxin-haemagglutinin complex (abobotulinumtoxinA).
- Placebo: Subjects received i.m. injections of placebo into the soleus muscle and gastrocnemius (medial and/or lateral) muscle and at least one of the distal or proximal muscles of the leg on Day 1 of the single treatment cycle.
Period: Overall Study
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Started | 127 | 129 | 132
Completed | 120 | 121 | 125
Not Completed | 7 | 8 | 7
Not completed — Study treatment not received | 0 | 1 | 2
Not completed — No MAS Score at baseline and/or Week 4 | 2 | 0 | 2
Not completed — Adverse Event | 2 | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2 | 0
Not completed — Botulinum toxin (BTX) in upper limb | 1 | 2 | 1
Not completed — Non compliance to visit schedule | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The ITT population included all randomised subjects who received at least 1 injection of study medication and who had a Modified Ashworth Scale (MAS) score in the gastrocnemius-soleus (GSC) assessed at baseline (pre-treatment) and at Week 4.
Groups:
- Dysport® 1000 U: Subjects received i.m.injections of Dysport® 1000 Units (U) (maximum total dose) into the soleus muscle and gastrocnemius (medial and/or lateral) muscle and at least one of the distal or proximal muscles of the leg on Day 1 of the single treatment cycle. Dysport® contains the neurotoxin Clostridium botulinum type A toxin-haemagglutinin complex (abobotulinumtoxinA).
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo | Total Title
Number analyzed (Participants) | 125 | 128 | 128 | 381
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (13.2) | 53.3 (12.0) | 51.4 (12.9) | 52.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 49 | 38 | 125
  Male | 87 | 79 | 90 | 256
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 4 | 3 | 10
  Black or African American | 5 | 13 | 5 | 23
  Caucasian or White | 116 | 109 | 119 | 344
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Multiple | 1 | 1 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 11 | 11 | 36
  Not Hispanic or Latino | 111 | 117 | 117 | 345

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Change From Baseline to Week 4 in the MAS Score in the Gastrocnemius-soleus Complex (GSC) (Knee Extended)
Description: Muscle tone in the treated limb was assessed by MAS in the GSC (with the knee extended) at baseline, at Weeks 1, 4 and 12, at discretionary visits at Weeks 16, 20 and 24, and at end of study. The MAS consists of 6 grades: 0 (no increase in muscle tone), 1 (slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion (ROM)), 1+ (slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM), 2 (more marked increase in muscle tone), 3 (considerable increase in muscle tone) or 4 (affected part(s) rigid in flexion or extension), and can be applied to muscles of both the upper and lower limbs. The least squares mean change from baseline at Week 4 is reported.
Time Frame: Baseline and Week 4
Population: The ITT population included all randomised subjects who received at least 1 injection of study medication and who had a MAS score in the GSC assessed at baseline (pre-treatment) and at Week 4.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Dysport® 1000 U: Subjects received i.m. injections of Dysport® 1000 Units (U) (maximum total dose) into the soleus muscle and gastrocnemius (medial and/or lateral) muscle and at least one of the distal or proximal muscles of the leg on Day 1 of the single treatment cycle. Dysport® contains the neurotoxin Clostridium botulinum type A toxin-haemagglutinin complex (abobotulinumtoxinA).
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 125 | 128 | 128
units on a scale | -0.6 [-0.8 to -0.5] | -0.8 [-0.9 to -0.7] | -0.5 [-0.7 to -0.4]
Statistical Analysis 1: Comparison: Dysport® 1000 U vs Placebo; The least squares mean change from baseline to Week 4 for MAS in the Dysport® 1000 U and Placebo groups were compared using 2 contrast analyses within a single mixed effect analysis of covariance (ANCOVA) model, controlling for the baseline values, the randomisation stratification factor (BTX treatment status at baseline) and the centre, all as fixed effects; Test type: Superiority or Other; p = 0.2859, ANCOVA; Least squares (LS) mean difference = -0.1, 95% CI 2-sided [-0.3 to 0.1] — LS Means for each treatment group and treatment comparisons as well as the p-values are obtained from an ANCOVA on the change from baseline with treatment, baseline MAS score, BTX treatment status at baseline and centre as covariates
Statistical Analysis 2: Comparison: Dysport® 1500 U vs Placebo; The least squares mean change from baseline to Week 4 for MAS in the Dysport® 1500 U and Placebo groups were compared using 2 contrast analyses within a single mixed effect ANCOVA model, controlling for the baseline values, the randomisation stratification factor (BTX treatment status at baseline) and the centre, all as fixed effects; Test type: Superiority or Other; p = 0.0091, ANCOVA; LS mean difference = -0.3, 95% CI 2-sided [-0.5 to -0.1] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Physician's Global Assesment (PGA) of Treatment Response at Week 4
Description: An assessment of overall treatment response was conducted at Weeks 4 and 12, and discretionary visits at Weeks 16, 20 and 24 and at end of study by an investigator who had not assessed the MAS. The investigator rated the response to treatment in the subject's lower limb after injection of Dysport® relative to the status at the baseline. Answers were made on a 9 point rating scale: -4=markedly worse, -3=much worse, -2=worse, -1=slightly worse, 0=no change, +1=slightly improved, +2=improved, +3=much improved, +4=markedly improved. The mean PGA score at Week 4 is reported.
Time Frame: At Week 4
Population: The ITT population included all randomised subjects who received at least 1 injection of study medication and who had a MAS score in the GSC assessed at baseline (pre-treatment) and at Week 4. Only subjects with data at Week 4 are included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 124 | 125 | 128
units on a scale | 0.9 [0.7 to 1.1] | 0.9 [0.7 to 1.1] | 0.7 [0.5 to 0.9]
Statistical Analysis 1: Comparison: Dysport® 1000 U vs Placebo; The mean PGA at Week 4 in the Dysport® 1000 U and Placebo groups were compared using 2 contrast analyses within a single mixed effect ANCOVA model, controlling for the baseline values, the randomisation stratification factor (BTX treatment status at baseline) and the centre, all as fixed effects; Test type: Superiority or Other; p = 0.0640, ANCOVA; LS mean difference = 0.3, 95% CI 2-sided [-0.0 to 0.5] — LS means for each treatment group and treatment comparisons as well as the p-values are obtained from an ANCOVA on visit results with treatment, BTX treatment status at baseline and centre as covariates
Statistical Analysis 2: Comparison: Dysport® 1500 U vs Placebo; The mean PGA at Week 4 in the Dysport® 1500 U and Placebo groups were compared using 2 contrast analyses within a single mixed effect ANCOVA model, controlling for the baseline values, the randomisation stratification factor (BTX treatment status at baseline) and the centre, all as fixed effects; Test type: Superiority or Other; p = 0.0665, ANCOVA; LS mean difference = 0.3, 95% CI 2-sided [-0.0 to 0.5] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Dysport® 1000 U vs Placebo; The LS mean rank values were back transformed to the original scale to give ranked PGA scores in an attempt to better normalise the data and restore power; Test type: Superiority or Other; p = 0.0466, ANCOVA on rank PGA scores; LS mean difference = 0.2 — LS means for each treatment group and treatment comparisons and the p-values are obtained from an analysis of variance on visit results based on ranked values with treatment, BTX treatment status at baseline and centre as explanatory variables
Statistical Analysis 4: Comparison: Dysport® 1500 U vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0406, ANCOVA on rank PGA scores; LS mean difference = 0.2 — [estimate comment as in outcome 2, analysis 3]

3. Secondary Outcome: Least Squares Mean Change From Baseline to Week 4 in Comfortable Barefoot Walking Speed
Description: Comfortable walking speed was assessed as a measure of functional ability and gait over 10 metres. Evaluations were made barefoot, without walking aids, at baseline and Weeks 1, 4 and 12 and discretionary visits at Weeks 16, 20 and 24 and at end of study. The least squares mean change from baseline at Week 4 is reported.
Time Frame: Baseline and Week 4
Population: The ITT population included all randomised subjects who received at least 1 injection of study medication and who had a MAS score in the GSC assessed at baseline (pre-treatment) and at Week 4. Only subjects with data at baseline and Week 4 are included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: m/s
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 124 | 127 | 126
m/s | 0.05 [0.03 to 0.07] | 0.04 [0.03 to 0.06] | 0.05 [0.03 to 0.07]
Statistical Analysis 1: Comparison: Dysport® 1000 U vs Placebo; The least squares mean change from baseline to Week 4 for barefoot comfortable walking speed in the Dysport® 1000 U and Placebo groups were compared using 2 contrast analyses within a single mixed effect analysis of covariance (ANCOVA) model, controlling for the baseline values, the randomisation stratification factor (BTX treatment status at baseline) and the centre, all as fixed effects; Test type: Superiority or Other; p = 0.7247, ANCOVA; LS mean difference = 0.01, 95% CI 2-sided [-0.02 to 0.03] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Dysport® 1500 U vs Placebo; The least squares mean change from baseline to Week 4 for barefoot comfortable walking speed in the Dysport® 1500 U and Placebo groups were compared using 2 contrast analyses within a single mixed effect ANCOVA model, controlling for the baseline values, the randomisation stratification factor (BTX treatment status at baseline) and the centre, all as fixed effects; Test type: Superiority or Other; p = 0.7266, ANCOVA; LS mean difference = -0.01, 95% CI 2-sided [-0.03 to 0.02] — [estimate comment as in outcome 1, analysis 1]

4. Other Pre Specified Outcome: Least Squares Mean Change From Baseline in MAS Score in the GSC (Knee Extended) at Weeks 1 and 12
Description: Muscle tone in the treated limb was assessed by MAS in the GSC (with the knee extended) at baseline, at Weeks 1, 4 and 12, at discretionary visits at Weeks 16, 20 and 24, and at end of study. The MAS consists of 6 grades: 0 (no increase in muscle tone), 1 (slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the ROM), 1+ (slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM), 2 (more marked increase in muscle tone), 3 (considerable increase in muscle tone) or 4 (affected part(s) rigid in flexion or extension), and can be applied to muscles of both the upper and lower limbs. The least squares mean change from baseline at Weeks 1 and 12 are reported.
Time Frame: Baseline and Weeks 1 and 12
Population: The ITT population included all randomised subjects who received at least 1 injection of study medication and who had a MAS score in the GSC assessed at baseline (pre-treatment) and at Week 4. Only subjects with data available at each timepoint presented are included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 125 | 128 | 128
units on a scale
  Week 1: number analyzed (Participants) | 123 | 128 | 128
  Week 1 | -0.4 [-0.6 to -0.3] | -0.5 [-0.6 to -0.4] | -0.4 [-0.5 to -0.2]
  Week 12: number analyzed (Participants) | 120 | 123 | 122
  Week 12 | -0.4 [-0.5 to -0.2] | -0.6 [-0.7 to -0.4] | -0.4 [-0.5 to -0.2]

5. Other Pre Specified Outcome: Least Squares Mean Change From Baseline in MAS Score in the Soleus (Knee Flexed) at Weeks 1, 4 and 12
Description: Muscle tone in the treated limb was assessed by MAS in the soleus (with the knee flexed) at baseline, at Weeks 1, 4 and 12, at discretionary visits at Weeks 16, 20 and 24, and at end of study. The MAS consists of 6 grades: 0 (no increase in muscle tone), 1 (slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the ROM), 1+ (slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM), 2 (more marked increase in muscle tone), 3 (considerable increase in muscle tone) or 4 (affected part(s) rigid in flexion or extension), and can be applied to muscles of both the upper and lower limbs. The least squares mean change from baseline at Weeks 1, 4 and 12 are reported.
Time Frame: Baseline and Weeks 1, 4 and 12
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 125 | 128 | 128
units on a scale
  Week 1: number analyzed (Participants) | 123 | 128 | 128
  Week 1 | -0.4 [-0.5 to -0.2] | -0.6 [-0.7 to -0.4] | -0.4 [-0.6 to -0.3]
  Week 4 | -0.7 [-0.8 to -0.5] | -0.8 [-1.0 to -0.7] | -0.4 [-0.6 to -0.3]
  Week 12: number analyzed (Participants) | 120 | 123 | 122
  Week 12 | -0.5 [-0.7 to -0.4] | -0.6 [-0.7 to -0.4] | -0.3 [-0.4 to -0.1]

6. Other Pre Specified Outcome: PGA of Treatment Response at Week 12
Description: An assessment of overall treatment response was conducted at Weeks 4 and 12, and discretionary visits at Weeks 16, 20 and 24 and at end of study by an investigator who had not assessed the MAS. The investigator rated the response to treatment in the subject's lower limb after injection of Dysport® relative to the status at the baseline. Answers were made on a 9 point rating scale: -4=markedly worse, -3=much worse, -2=worse, -1=slightly worse, 0=no change, +1=slightly improved, +2=improved, +3=much improved, +4=markedly improved. The mean PGA scores at Week 12 are reported.
Time Frame: At Week 12
Population: The ITT population included all randomised subjects who received at least 1 injection of study medication and who had a MAS score in the GSC assessed at baseline (pre-treatment) and at Week 4. Only subjects with data at Week 12 are included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 120 | 123 | 122
units on a scale | 0.6 [0.4 to 0.7] | 0.6 [0.4 to 0.8] | 0.5 [0.3 to 0.7]

7. Other Pre Specified Outcome: Least Squares Mean Change From Baseline in Comfortable Barefoot Walking Speed at Weeks 1 and 12
Description: Comfortable walking speed was assessed as a measure of functional ability and gait over 10 metres. Evaluations were made barefoot, without walking aids, at baseline and Weeks 1, 4 and 12 and discretionary visits at Weeks 16, 20 and 24 and at end of study. The least squares mean change from baseline at Weeks 1 and 12 are reported.
Time Frame: Baseline and Weeks 1 and 12
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: m/s
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 125 | 128 | 128
m/s
  Week 1: number analyzed (Participants) | 123 | 127 | 127
  Week 1 | 0.05 [0.04 to 0.07] | 0.04 [0.02 to 0.05] | 0.04 [0.02 to 0.05]
  Week 12: number analyzed (Participants) | 120 | 120 | 120
  Week 12 | 0.07 [0.05 to 0.09] | 0.06 [0.04 to 0.08] | 0.05 [0.03 to 0.07]

8. Other Pre Specified Outcome: Least Squares Mean Change From Baseline in Comfortable Walking Speed With Shoes at Weeks 1, 4 and 12
Description: Comfortable walking speed was assessed as a measure of functional ability and gait over 10 metres. Evaluations were made with shoes, without walking aids, at baseline and Weeks 1, 4 and 12 and discretionary visits at Weeks 16, 20 and 24 and at end of study. The least squares mean change from baseline at Weeks 1, 4 and 12 are reported.
Time Frame: Baseline and Weeks 1, 4 and 12
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: m/s
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 125 | 128 | 128
m/s
  Week 1: number analyzed (Participants) | 122 | 127 | 127
  Week 1 | 0.05 [0.03 to 0.07] | 0.05 [0.03 to 0.07] | 0.04 [0.02 to 0.05]
  Week 4: number analyzed (Participants) | 124 | 127 | 127
  Week 4 | 0.05 [0.03 to 0.07] | 0.04 [0.02 to 0.06] | 0.06 [0.04 to 0.08]
  Week 12: number analyzed (Participants) | 119 | 121 | 122
  Week 12 | 0.06 [0.04 to 0.08] | 0.05 [0.03 to 0.07] | 0.05 [0.03 to 0.07]

9. Other Pre Specified Outcome: Least Squares Mean Change From Baseline in Maximal Barefoot Walking Speed at Weeks 1, 4 and 12
Description: Maximal walking speed was assessed as a measure of functional ability and gait over 10 metres. Evaluations were made barefoot, without walking aids, at baseline and Weeks 1, 4 and 12 and discretionary visits at Weeks 16, 20 and 24 and at end of study. The least squares mean change from baseline at Weeks 1, 4 and are reported.
Time Frame: Baseline and Weeks 1, 4 and 12
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: m/s
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 125 | 128 | 128
m/s
  Week 1: number analyzed (Participants) | 123 | 127 | 127
  Week 1 | 0.06 [0.04 to 0.08] | 0.05 [0.03 to 0.07] | 0.05 [0.03 to 0.07]
  Week 4: number analyzed (Participants) | 124 | 127 | 125
  Week 4 | 0.07 [0.05 to 0.10] | 0.04 [0.02 to 0.06] | 0.05 [0.03 to 0.08]
  Week 12: number analyzed (Participants) | 120 | 120 | 120
  Week 12 | 0.09 [0.06 to 0.12] | 0.06 [0.03 to 0.08] | 0.06 [0.03 to 0.09]

10. Other Pre Specified Outcome: Least Squares Mean Change From Baseline in Maximal Walking Speed With Shoes at Weeks 1, 4 and 12
Description: Maximal walking speed was assessed as a measure of functional ability and gait over 10 metres. Evaluations were made with shoes, without walking aids, at baseline and Weeks 1, 4 and 12 and discretionary visits at Weeks 16, 20 and 24 and at end of study. The least squares mean change from baseline at Weeks 1, 4 and 12 are reported.
Time Frame: Baseline and Weeks 1, 4 and 12
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: m/s
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 125 | 128 | 128
m/s
  Week 1: number analyzed (Participants) | 121 | 127 | 127
  Week 1 | 0.05 [0.03 to 0.07] | 0.05 [0.03 to 0.07] | 0.04 [0.03 to 0.06]
  Week 4: number analyzed (Participants) | 123 | 127 | 127
  Week 4 | 0.05 [0.03 to 0.08] | 0.04 [0.02 to 0.07] | 0.05 [0.03 to 0.08]
  Week 12: number analyzed (Participants) | 118 | 121 | 122
  Week 12 | 0.07 [0.04 to 0.10] | 0.05 [0.03 to 0.08] | 0.05 [0.02 to 0.08]

11. Other Pre Specified Outcome: Least Squares Mean Change From Baseline in Cadence With Comfortable Walking Speed With Shoes at Weeks 1, 4 and 12
Description: Cadence was assessed during the 10-metre walking speed test at comfortable walking speed and with shoes. The evaluator walked beside the subject during the test and counted the number of steps taken during the 10-metre walk. The gait parameters were measured at baseline, Weeks 1, 4 and 12, discretionary visits at Weeks 16, 20 and 24 and at end of study. The least squares mean change from baseline at Weeks 1, 4 and 12 are reported.
Time Frame: Baseline and Weeks 1, 4 and 12
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: steps/s
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 125 | 128 | 128
steps/s
  Week 1: number analyzed (Participants) | 122 | 127 | 127
  Week 1 | 0.07 [0.04 to 0.10] | 0.07 [0.04 to 0.10] | 0.04 [0.01 to 0.07]
  Week 4: number analyzed (Participants) | 124 | 127 | 127
  Week 4 | 0.07 [0.04 to 0.10] | 0.06 [0.03 to 0.10] | 0.06 [0.02 to 0.09]
  Week 12: number analyzed (Participants) | 119 | 121 | 122
  Week 12 | 0.09 [0.05 to 0.12] | 0.06 [0.03 to 0.09] | 0.05 [0.01 to 0.08]

12. Other Pre Specified Outcome: Least Squares Mean Change From Baseline in Average Step Length With Comfortable Walking Speed With Shoes at Weeks 1, 4 and 12
Description: Average step length was assessed during the 10-metre walking speed test at comfortable walking speed and with shoes. The evaluator walked beside the subject during the test and counted the number of steps taken during the 10-metre walk. The gait parameters were measured at baseline, Weeks 1, 4 and 12, discretionary visits at Weeks 16, 20 and 24 and at end of study. The least squares mean change from baseline at Weeks 1, 4 and 12 are reported.
Time Frame: Baseline and Weeks 1, 4 and 12
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: m/step
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 125 | 128 | 128
m/step
  Week 1: number analyzed (Participants) | 122 | 127 | 127
  Week 1 | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.03]
  Week 4: number analyzed (Participants) | 124 | 127 | 127
  Week 4 | 0.02 [0.01 to 0.03] | 0.01 [0.0 to 0.02] | 0.03 [0.02 to 0.04]
  Week 12: number analyzed (Participants) | 119 | 121 | 122
  Week 12 | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.04] | 0.03 [0.01 to 0.04]

13. Other Pre Specified Outcome: Least Squares Mean Change From Baseline in Cadence With Comfortable Barefoot Walking Speed at Weeks 1, 4 and 12
Description: Cadence was assessed during the 10-metre walking speed test at comfortable walking speed and barefoot. The evaluator walked beside the subject during the test and counted the number of steps taken during the 10-metre walk. The gait parameters were measured at baseline, Weeks 1, 4 and 12, discretionary visits at Weeks 16, 20 and 24 and at end of study. The least squares mean change from baseline at Weeks 1, 4 and 12 are reported
Time Frame: Baseline and Weeks 1, 4 and 12
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: steps/s
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 125 | 128 | 128
steps/s
  Week 1: number analyzed (Participants) | 123 | 127 | 127
  Week 1 | 0.10 [0.07 to 0.13] | 0.05 [0.02 to 0.08] | 0.05 [0.02 to 0.08]
  Week 4: number analyzed (Participants) | 124 | 127 | 126
  Week 4 | 0.08 [0.04 to 0.11] | 0.06 [0.03 to 0.10] | 0.06 [0.02 to 0.09]
  Week 12: number analyzed (Participants) | 120 | 120 | 120
  Week 12 | 0.12 [0.08 to 0.15] | 0.08 [0.05 to 0.12] | 0.07 [0.04 to 0.11]

14. Other Pre Specified Outcome: Least Squares Mean Change From Baseline in Average Step Length With Comfortable Barefoot Walking Speed at Weeks 1, 4 and 12
Description: Average step length was assessed during the 10-metre walking speed test at comfortable walking speed and barefoot. The evaluator walked beside the subject during the test and counted the number of steps taken during the 10-metre walk. The gait parameters were measured at baseline, Weeks 1, 4 and 12, discretionary visits at Weeks 16, 20 and 24 and at end of study. The least squares mean change from baseline at Weeks 1, 4 and 12 are reported.
Time Frame: Baseline and Weeks 1, 4 and 12
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: m/step
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 125 | 128 | 128
m/step
  Week 1: number analyzed (Participants) | 123 | 127 | 127
  Week 1 | 0.02 [0.01 to 0.02] | 0.02 [0.01 to 0.02] | 0.01 [0.00 to 0.02]
  Week 4: number analyzed (Participants) | 124 | 127 | 126
  Week 4 | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.03]
  Week 12: number analyzed (Participants) | 120 | 120 | 120
  Week 12 | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.03]

15. Other Pre Specified Outcome: Least Squares Mean Change From Baseline in Cadence With Maximal Walking Speed With Shoes at Weeks 1, 4 and 12
Description: Cadence was assessed during the 10-metre walking speed test at maximal walking speed and with shoes. The evaluator walked beside the subject during the test and counted the number of steps taken during the 10-metre walk. The gait parameters were measured at baseline, Weeks 1, 4 and 12, discretionary visits at Weeks 16, 20 and 24 and at end of study. The least squares mean change from baseline at Weeks 1, 4 and 12 are reported.
Time Frame: Baseline and Weeks 1, 4 and 12
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: steps/s
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 125 | 128 | 128
steps/s
  Week 1: number analyzed (Participants) | 121 | 127 | 127
  Week 1 | 0.06 [0.02 to 0.09] | 0.07 [0.03 to 0.10] | 0.04 [0.01 to 0.08]
  Week 4: number analyzed (Participants) | 123 | 127 | 127
  Week 4 | 0.05 [0.02 to 0.09] | 0.05 [0.02 to 0.09] | 0.05 [0.02 to 0.09]
  Week 12: number analyzed (Participants) | 118 | 121 | 122
  Week 12 | 0.08 [0.04 to 0.12] | 0.07 [0.03 to 0.11] | 0.04 [-0.00 to 0.08]

16. Other Pre Specified Outcome: Least Squares Mean Change From Baseline in Average Step Length With Maximal Walking Speed With Shoes at Weeks 1, 4 and 12
Description: Average step length was assessed during the 10-metre walking speed test at maximal walking speed and with shoes. The evaluator walked beside the subject during the test and counted the number of steps taken during the 10-metre walk. The gait parameters were measured at baseline, Weeks 1, 4 and 12, discretionary visits at Weeks 16, 20 and 24 and at end of study. The least squares mean change from baseline at Weeks 1, 4 and 12 are reported.
Time Frame: Baseline and Weeks 1, 4 and 12
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: m/step
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 125 | 128 | 128
m/step
  Week 1: number analyzed (Participants) | 121 | 127 | 127
  Week 1 | 0.02 [0.00 to 0.03] | 0.01 [0.00 to 0.03] | 0.02 [0.01 to 0.04]
  Week 4: number analyzed (Participants) | 123 | 127 | 127
  Week 4 | 0.02 [0.00 to 0.03] | 0.02 [0.00 to 0.03] | 0.02 [0.01 to 0.03]
  Week 12: number analyzed (Participants) | 118 | 121 | 122
  Week 12 | 0.02 [0.00 to 0.03] | 0.02 [0.00 to 0.03] | 0.03 [0.01 to 0.04]

17. Other Pre Specified Outcome: Least Squares Mean Change From Baseline in Cadence With Maximal Barefoot Walking Speed at Weeks 1, 4 and 12
Description: Cadence was assessed during the 10-metre walking speed test at maximal walking speed and barefoot. The evaluator walked beside the subject during the test and counted the number of steps taken during the 10-metre walk. The gait parameters were measured at baseline, Weeks 1, 4 and 12, discretionary visits at Weeks 16, 20 and 24 and at end of study. The least squares mean change from baseline at Weeks 1, 4 and 12 are reported.
Time Frame: Baseline and Weeks 1, 4 and 12
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: steps/s
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 125 | 128 | 128
steps/s
  Week 1: number analyzed (Participants) | 123 | 127 | 127
  Week 1 | 0.07 [0.04 to 0.11] | 0.05 [0.02 to 0.09] | 0.06 [0.02 to 0.09]
  Week 4: number analyzed (Participants) | 124 | 127 | 125
  Week 4 | 0.08 [0.04 to 0.12] | 0.05 [0.01 to 0.09] | 0.07 [0.03 to 0.10]
  Week 12: number analyzed (Participants) | 120 | 120 | 120
  Week 12 | 0.12 [0.08 to 0.16] | 0.08 [0.03 to 0.12] | 0.06 [0.02 to 0.11]

18. Other Pre Specified Outcome: Least Squares Mean Change From Baseline in Average Step Length With Maximal Barefoot Walking Speed at Weeks 1, 4 and 12
Description: Average step length was assessed during the 10-metre walking speed test at maximal walking speed and barefoot. The evaluator walked beside the subject during the test and counted the number of steps taken during the 10-metre walk. The gait parameters were measured at baseline, Weeks 1, 4 and 12, discretionary visits at Weeks 16, 20 and 24 and at end of study. The least squares mean change from baseline at Weeks 1, 4 and 12 are reported.
Time Frame: Baseline and Weeks 1, 4 and 12
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: m/step
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 125 | 128 | 128
m/step
  Week 1: number analyzed (Participants) | 123 | 127 | 127
  Week 1 | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.03]
  Week 4: number analyzed (Participants) | 124 | 127 | 125
  Week 4 | 0.02 [0.01 to 0.04] | 0.02 [0.00 to 0.03] | 0.02 [0.00 to 0.03]
  Week 12: number analyzed (Participants) | 120 | 120 | 120
  Week 12 | 0.02 [0.01 to 0.03] | 0.02 [0.00 to 0.03] | 0.02 [0.01 to 0.04]

19. Other Pre Specified Outcome: Least Squares Mean Change From Baseline in the Tardieu Scale in the GSC (Knee Extended) at Weeks 1, 4 and 12: Angle of Arrest (XV1), Angle of Catch (XV3) and Spasticity Angle (X)
Description: The Tardieu Scale in the GSC was used to assess spasticity with the knee extended. Assessments were made at slow (V1) and fast (V3) speeds of stretch. Slow speed of muscle stretch measures the range of passive motion. During a slow stretching movement, the examiner determines the angle of movement arrest (XV1), either due to subject discomfort or a mechanical resistance. The same movement is repeated at a fast speed to determine the angle of catch and release (XV3). The spasticity angle (X) was calculated as the difference between XV1 and XV3. The Tardieu Scale ratings were made prior to the study treatment at baseline, and then after injection at Weeks 1, 4 and 12, and at discretionary visits if required at Weeks 16, 20 and 24 and at end of study. The least squares mean change from baseline at Weeks 1, 4 and 12 are reported.
Time Frame: Baseline and Weeks 1, 4 and 12
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Degrees
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 125 | 128 | 128
Degrees
  Week 1: Angle of Arrest (XV1): number analyzed (Participants) | 123 | 127 | 128
  Week 1: Angle of Arrest (XV1) | 2.4 [1.4 to 3.4] | 2.3 [1.3 to 3.3] | 1.7 [0.7 to 2.6]
  Week 4: Angle of Arrest (XV1): number analyzed (Participants) | 125 | 128 | 127
  Week 4: Angle of Arrest (XV1) | 0.7 [-0.5 to 1.9] | 1.4 [0.2 to 2.6] | 1.3 [0.1 to 2.5]
  Week 12: Angle of Arrest (XV1): number analyzed (Participants) | 120 | 123 | 122
  Week 12: Angle of Arrest (XV1) | 0.4 [-0.9 to 1.7] | 0.4 [-0.9 to 1.6] | 0.5 [-0.8 to 1.7]
  Week 1: Angle of Catch (XV3): number analyzed (Participants) | 123 | 128 | 128
  Week 1: Angle of Catch (XV3) | 5.1 [3.8 to 6.5] | 5.4 [4.1 to 6.7] | 3.2 [1.9 to 4.5]
  Week 4: Angle of Catch (XV3) | 4.8 [3.3 to 6.3] | 5.3 [3.8 to 6.8] | 3.4 [1.9 to 4.9]
  Week 12: Angle of Catch (XV3): number analyzed (Participants) | 120 | 123 | 122
  Week 12: Angle of Catch (XV3) | 3.0 [1.4 to 4.6] | 2.9 [1.3 to 4.5] | 2.6 [1.0 to 4.2]
  Week 1: Spasticity Angle (X): number analyzed (Participants) | 123 | 127 | 128
  Week 1: Spasticity Angle (X) | -2.5 [-3.7 to -1.3] | -3.2 [-4.4 to -2.0] | -1.7 [-2.8 to -0.5]
  Week 4: Spasticity Angle (X): number analyzed (Participants) | 125 | 128 | 127
  Week 4: Spasticity Angle (X) | -4.0 [-5.2 to -2.8] | -4.0 [-5.2 to -2.8] | -2.5 [-3.7 to -1.3]
  Week 12: Spasticity Angle (X): number analyzed (Participants) | 120 | 123 | 122
  Week 12: Spasticity Angle (X) | -2.4 [-3.7 to -1.1] | -2.8 [-4.0 to -1.5] | -2.3 [-3.5 to -1.0]

20. Other Pre Specified Outcome: Least Squares Mean Change From Baseline in the Tardieu Scale in the GSC (Knee Extended) at Weeks 1, 4 and 12: Spasticity Grade (Y)
Description: The Tardieu Scale in the GSC was used to assess spasticity with the knee extended. The spasticity grade (Y) assesses quality of muscle reaction on a 5-point scale (measured at fast speed): 0 = no resistance throughout passive movement; 1 = slight resistance throughout passive movement; 2 = clear catch at precise angle, interrupting passive movement, followed by release; 3 = fatigable clonus (less than 10 seconds when maintaining pressure) occurring at a precise angle, followed by release; 4 = unfatigable clonus (more than 10 seconds when maintaining pressure) occurring at precise angle. The Tardieu Scale ratings were made prior to the study treatment at baseline, and then after injection at Weeks 1, 4 and 12, and at discretionary visits if required at Weeks 16, 20 and 24 and at end of study. The least squares mean change from baseline for spasticity grade at Weeks 1, 4 and 12 are reported.
Time Frame: Baseline and Weeks 1, 4 and 12
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 125 | 128 | 128
units on a scale
  Week 1: number analyzed (Participants) | 123 | 127 | 128
  Week 1 | -0.2 [-0.3 to -0.1] | -0.3 [-0.4 to -0.2] | -0.2 [-0.3 to -0.1]
  Week 4 | -0.3 [-0.4 to -0.2] | -0.4 [-0.5 to -0.3] | -0.1 [-0.2 to -0.0]
  Week 12: number analyzed (Participants) | 120 | 123 | 122
  Week 12 | -0.3 [-0.4 to -0.2] | -0.4 [-0.5 to -0.3] | -0.1 [-0.2 to -0.0]

21. Other Pre Specified Outcome: Least Squares Mean Change From Baseline in the Tardieu Scale in the Soleus (Knee Flexed) at Weeks 1, 4 and 12: Angle of Arrest (XV1), Angle of Catch (XV3) and Spasticity Angle (X)
Description: The Tardieu Scale in the soleus was used to assess spasticity with the knee flexed. Assessments were made at slow (V1) and fast (V3) speeds of stretch. Slow speed of muscle stretch measures the range of passive motion. During a slow stretching movement, the examiner determines the angle of movement arrest (XV1), either due to subject discomfort or a mechanical resistance. The same movement is repeated at a fast speed to determine the angle of catch and release (XV3). The spasticity angle (X) was calculated as the difference between XV1 and XV3. The Tardieu Scale ratings were made prior to the study treatment at baseline, and then after injection at Weeks 1, 4 and 12, and at discretionary visits if required at Weeks 16, 20 and 24 and at end of study. The least squares mean change from baseline at Weeks 1, 4 and 12 are reported.
Time Frame: Baseline and Weeks 1, 4 and 12
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Degrees
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 125 | 128 | 128
Degrees
  Week 1: Angle of Arrest (XV1): number analyzed (Participants) | 123 | 127 | 128
  Week 1: Angle of Arrest (XV1) | 2.2 [1.2 to 3.2] | 1.5 [0.6 to 2.5] | 1.4 [0.4 to 2.3]
  Week 4: Angle of Arrest (XV1) | 1.2 [0.1 to 2.3] | 1.0 [-0.1 to 2.1] | 1.3 [0.2 to 2.4]
  Week 12: Angle of Arrest (XV1): number analyzed (Participants) | 120 | 123 | 122
  Week 12: Angle of Arrest (XV1) | 0.4 [-0.7 to 1.5] | 0.1 [-1.0 to 1.1] | 0.0 [-1.0 to 1.1]
  Week 1: Angle of Catch (XV3): number analyzed (Participants) | 123 | 128 | 128
  Week 1: Angle of Catch (XV3) | 4.1 [2.5 to 5.8] | 4.1 [2.5 to 5.8] | 2.5 [0.9 to 4.1]
  Week 4: Angle of Catch (XV3) | 5.1 [3.5 to 6.6] | 4.9 [3.4 to 6.4] | 2.9 [1.5 to 4.4]
  Week 12: Angle of Catch (XV3): number analyzed (Participants) | 120 | 123 | 122
  Week 12: Angle of Catch (XV3) | 4.0 [2.5 to 5.4] | 3.7 [2.2 to 5.1] | 2.7 [1.2 to 4.1]
  Week 1: Spasticity Angle (X): number analyzed (Participants) | 123 | 127 | 128
  Week 1: Spasticity Angle (X) | -1.7 [-3.1 to -0.2] | -2.8 [-4.2 to -1.4] | -1.3 [-2.6 to -0.1]
  Week 4: Spasticity Angle (X) | -3.6 [-4.9 to -2.4] | -4.2 [-5.5 to -3.0] | -1.8 [-3.1 to -0.6]
  Week 12: Spasticity Angle (X): number analyzed (Participants) | 120 | 123 | 122
  Week 12: Spasticity Angle (X) | -3.3 [-4.6 to -2.1] | -3.9 [-5.2 to -2.7] | -2.8 [-4.1 to -1.6]

22. Other Pre Specified Outcome: Least Squares Mean Change From Baseline in the Tardieu Scale in the Soleus (Knee Flexed) at Weeks 1, 4 and 12: Spasticity Grade (Y)
Description: The Tardieu Scale in the soleus was used to assess spasticity with the knee flexed. The spasticity grade (Y) assesses quality of muscle reaction on a 5-point scale (measured at fast speed): 0 = no resistance throughout passive movement; 1 = slight resistance throughout passive movement; 2 = clear catch at precise angle, interrupting passive movement, followed by release; 3 = fatigable clonus (less than 10 seconds when maintaining pressure) occurring at a precise angle, followed by release; 4 = unfatigable clonus (more than 10 seconds when maintaining pressure) occurring at precise angle. The Tardieu Scale ratings were made prior to the study treatment at baseline, and then after injection at Weeks 1, 4 and 12, and at discretionary visits if required at Weeks 16, 20 and 24 and at end of study. The least squares mean change from baseline for spasticity grade at Weeks 1, 4 and 12 are reported.
Time Frame: Baseline and Weeks 1, 4 and 12
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 125 | 128 | 128
units on a scale
  Week 1: number analyzed (Participants) | 123 | 127 | 128
  Week 1 | -0.2 [-0.3 to -0.1] | -0.3 [-0.4 to -0.2] | -0.1 [-0.2 to -0.0]
  Week 4 | -0.5 [-0.6 to -0.3] | -0.5 [-0.6 to -0.4] | -0.1 [-0.2 to -0.0]
  Week 12: number analyzed (Participants) | 120 | 123 | 122
  Week 12 | -0.4 [-0.5 to -0.3] | -0.4 [-0.5 to -0.3] | -0.1 [-0.2 to -0.0]

23. Other Pre Specified Outcome: Least Squares Mean Change From Baseline in the Range of Active Dorsiflexion at Weeks 1, 4 and 12 (Knee Extended and Flexed)
Description: Range of active dorsiflexion of the ankle joint, both with the knee flexed (90°) and extended (measured by goniometry) was used to assess treatment response. The measurements were made prior to the study treatment at baseline, and then after injection at Weeks 1, 4 and 12, and at discretionary visits when needed at Weeks 16, 20 and 24 and at end of study. The least squares mean change from baseline at Weeks 1, 4 and 12 are reported.
Time Frame: Baseline and Weeks 1, 4 and 12
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Degrees
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 125 | 128 | 128
Degrees
  Week 1: Knee Extended: number analyzed (Participants) | 123 | 128 | 128
  Week 1: Knee Extended | 1.7 [0.4 to 3.0] | 2.4 [1.1 to 3.7] | 1.1 [-0.2 to 2.4]
  Week 4: Knee Extended: number analyzed (Participants) | 125 | 128 | 127
  Week 4: Knee Extended | 1.5 [-0.2 to 3.1] | 3.7 [2.0 to 5.3] | 1.6 [-0.1 to 3.2]
  Week 12: Knee Extended: number analyzed (Participants) | 119 | 123 | 122
  Week 12: Knee Extended | 1.1 [-0.5 to 2.7] | 2.0 [0.5 to 3.6] | 1.7 [0.1 to 3.2]
  Week 1: Knee Flexed: number analyzed (Participants) | 123 | 127 | 128
  Week 1: Knee Flexed | 3.0 [1.5 to 4.4] | 2.0 [0.6 to 3.4] | 1.9 [0.5 to 3.3]
  Week 4: Knee Flexed | 2.9 [1.4 to 4.5] | 3.3 [1.8 to 4.9] | 2.7 [1.2 to 4.2]
  Week 12: Knee Flexed: number analyzed (Participants) | 119 | 123 | 121
  Week 12: Knee Flexed | 2.0 [0.4 to 3.6] | 1.4 [-0.1 to 2.9] | 1.8 [0.2 to 3.3]

24. Other Pre Specified Outcome: Least Squares Mean Change From Baseline in Lower Limb Pain at Weeks 1, 4 and 12
Description: The intensity of lower limb pain was evaluated using the Scale of Pain Intensity (SPIN) which provided a pictorial representation of pain in a 6-point graphic scale with the degree of red shading inside a circle representing the intensity of pain. The bottom and top of the scale are anchored by two extremes: 'no pain' (circle with no red shading and scored as 0) and 'pain as bad as it could be' (circle completely red and scored as 5), marked with either verbal or visual cues. The intervening points are represented by red circles increasing proportionally in size. The subject marks the circle that best indicates their pain intensity. The SPIN assessments were obtained prior to the study treatment at baseline, and then after injection at Weeks 1, 4 and 12, and at discretionary visits when needed at Weeks 16, 20 and 24 and at end of study. The least squares mean change from baseline at Weeks 1, 4 and 12 are reported.
Time Frame: Baseline and Weeks 1, 4 and 12
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Number analyzed (Participants) | 125 | 128 | 128
units on a scale
  Week 1: number analyzed (Participants) | 121 | 127 | 128
  Week 1 | -0.3 [-0.4 to -0.1] | -0.1 [-0.3 to 0.0] | -0.2 [-0.3 to -0.0]
  Week 4: number analyzed (Participants) | 122 | 126 | 128
  Week 4 | -0.1 [-0.3 to -0.1] | -0.2 [-0.4 to 0.0] | -0.1 [-0.3 to 0.1]
  Week 12: number analyzed (Participants) | 118 | 121 | 122
  Week 12 | -0.2 [-0.4 to 0.0] | -0.1 [-0.3 to 0.1] | 0.1 [-0.1 to 0.3]

ADVERSE EVENTS:
Time Frame: From baseline up to Week 24 +/- 2 weeks.
Description: Adverse event (AE) data is reported as treatment emergent AEs; an AE was reported as emergent if it arose (i.e. started or worsened in severity) after the subject received study medication and were monitored from the time that the subject gave informed consent to the end of the study. All AEs were elicited by direct, non-leading questioning or by spontaneous reports. The safety population consisted of all randomised subjects who received at least 1 injection of study medication.
Arm/Group | Dysport® 1000 U | Dysport® 1500 U | Placebo
Serious Adverse Events (participants affected / at risk) | 5/127 | 5/128 | 7/130
Other Adverse Events (participants affected / at risk) | 22/127 | 21/128 | 11/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport® 1000 U (N=127) | Dysport® 1500 U (N=128) | Placebo (N=130)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) — Death (in placebo subject)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Death
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport® 1000 U (N=127) | Dysport® 1500 U (N=128) | Placebo (N=130)
Fall (Injury, poisoning and procedural complications) | 12 (14) | 8 (9) | 4 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 8 (9) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (8) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No